CLINICAL TRIAL: NCT01109745
Title: Effectiveness of the Paediatric Electronic Quality of Life Instrument for Childhood Asthma in the Netherlands (Pelican) in Medical Care.
Brief Title: Effectiveness of the Pelican Instrument in Medical Care
Acronym: PELICANII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, T. Schermer, PhD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NL29895.091.09; 3.4.07.043 (Other Grant/Funding Number: Dutch Asthma Foundation); 0802-74 (Other Grant/Funding Number: NutsOhra Foundation)
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: Asthma; health-related quality of life; patient-centred care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- usual primary care (No Intervention): Number of participating children: 85
- PELICAN Primary care (Experimental): Intervention arm: the integration of the output of the Pelican instrument (i.e., individualised HRQL information) in daily care to guide disease management for children with asthma treated in primary care. Number of participants: 85 children
  Interventions: Other: PELICAN Primary Care
- usual secondary care (No Intervention): number of participating children: 50
- PELICAN Secondary Care (Experimental): Intervention arm: the integration of the output of the Pelican instrument (i.e., individualised HRQL information) in daily care to guide disease management for children with asthma treated in primary care. Number of participants: 50 children
  Interventions: Other: PELICAN Secondary Care

INTERVENTIONS:
Other: PELICAN Primary Care — The intervention is the integration of the output of the Pelican instrument in daily care to guide disease management for children with asthma treated in primary care. The general practitioner can integrate the information of the Pelican instrument in their consultation and disease management decisions. The general practitioner will be trained and supported to negotiate the child's, and physicians' agendas based on the outcome of the instrument, and discuss possible interventions. All participating children of a GP will be allocated to the same treatment group (i.e., hierarchical or nested design).
  Arms: PELICAN Primary care
Other: PELICAN Secondary Care — The intervention is the integration of the output of the Pelican instrument in daily care to guide disease management for children with asthma treated in secondary care. The nurse can integrate the information of the Pelican instrument in their consultation and disease management decisions. The paediatricians will be trained and supported to negotiate the child's, and nurses' agendas based on the outcome of the instrument, and discuss possible interventions.
  Arms: PELICAN Secondary Care

SUMMARY:
The objective of this project is to establish the effectiveness of implementation of a self-administered electronic asthma-specific quality of life instrument for childhood asthma in primary care and specialist care.

DETAILED DESCRIPTION:
Health related quality of life (HRQL) is important to the asthmatic child and if HRQL aspects are taken into account in daily care this could result in improved treatment satisfaction, compliance, asthma control and, ultimately, improved HRQL. The Pelican instrument we have developed has the essential features to be useful in daily care. In this study, the effectiveness of implementing the Pelican instrument in medical care is assessed. An intervention study with 9 months follow-up in primary and secondary care will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* age 6 to 12 years
* physician-diagnosed asthma
* use of bronchodilators and / or inhaled corticosteroids for at least six weeks during the previous year
* child is treated for its asthma by the recruiting physician
* signed informed consent by parent (or caretaker)
* child agrees to participate in the study

Exclusion Criteria:

* comorbid condition that significantly influences HRQL
* child does not master the Dutch language sufficiently
* not being able to attend a regular school class

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
quality of life | 9 months
  Asthma specific health related quality of life measured with the Pediatric asthma quality of life questionnaire PAQLQ(S)

SECONDARY OUTCOMES:
asthma control | 9 months
  asthma control will be measured with the Asthma Control Questionnaire (ACQ) and the Childhood Asthma Control Test (C-ACT)
Symptoms and medication | 9 months
  asthmatic symptoms (e.g., wheezing, dyspnea) and medication use (e.g., use of inhaled corticosteroids, and short-acting bronchodilators) are assessed with a diary
Lung function | 9 months
  Lung function indices (FEV1 and FVC before and 15 minutes after inhalation of 400 µg salbutamol) are measured by a certified lung function technician specifically trained to coach children using a spirometer with child-incentive. Spirometry tests will be performed according to ERS/ATS spirometry standards and recommendations regarding testing in children. Spirometry is performed at least 8 hrs after the last inhalation of a short-acting bronchodilator, and 12 hrs after a long-acting bronchodilator.
Cost-effectiveness | 9 months
  A cost-effectiveness analysis (CEA) from a societal perspective will be performed and reported according to national and international guidelines. In the CEA an effect is defined as a relevant change in HRQL (i.e., ∆PAQLQ ≥0.5 point) in the denominator and the total of all relevant costs in the nominator. C/E ratios with and without inclusion of the indirect cost will be reported. A sensitivity analysis will be performed in order to estimate the susceptibility of C/E ratio's to variation in prior assumptions and choices, including 'worst case - best case' scenarios.
caregiver quality of life | 9 months
  The quality of life of the parents of the participating children is assessed with the Paediatric asthma caregiver quality of life (PACQoL) instrument.
process-outcomes | 9 months
  The implementation of the Pelican instrument in daily care is an complex intervention. A detailed process evaluation is crucial to evaluate how the intervention works: what are the active ingredients and how are they exerting their effect?

CONTACTS AND LOCATIONS:
Overall Officials: Lisette van den Bemt, PhD, Principal Investigator — Radboud University Medical Center; Tjard RJ Schermer, PhD, Study Director — Radboud University Medical Center
Locations (6):
- Netherlands (6):
  - Amphia Ziekenhuis, Breda, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Reinier de Graaf Groep, Delft, South Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Viecuri Medical Centre, Venlo

REFERENCES:
- [Background] van den Bemt L, Kooijman S, Linssen V, Lucassen P, Muris J, Slabbers G, Schermer T. How does asthma influence the daily life of children? Results of focus group interviews. Health Qual Life Outcomes. 2010 Jan 14;8:5. doi: 10.1186/1477-7525-8-5. PMID 20074334
- [Derived] van Bragt S, van den Bemt L, Cretier R, van Weel C, Merkus P, Schermer T. PELICAN: Content evaluation of patient-centered care for children with asthma based on an online tool. Pediatr Pulmonol. 2016 Oct;51(10):993-1003. doi: 10.1002/ppul.23397. Epub 2016 Apr 29. PMID 27128738
- [Derived] van Bragt S, van den Bemt L, Thoonen B, van Weel C, Merkus P, Schermer T. PELICAN: A quality of life instrument for childhood asthma: study protocol of two randomized controlled trials in primary and specialized care in the Netherlands. BMC Pediatr. 2012 Aug 30;12:137. doi: 10.1186/1471-2431-12-137. PMID 22935133
- See also: Website Radboud University Nijmegen Medical Centre (in Dutch) — http://www.umcn.nl
- See also: Website of the project for participants (in Dutch) — http://pelikaan.ruhosting.nl